CLINICAL TRIAL: NCT06861998
Title: The Impact of Behavioral Intervention On Postoperative Delirium In Sleep-Disordered Infants and Toddlers Undergoing Congenital Heart Surgery: A Multicenter, Randomized Controlled Clinical Trial
Brief Title: Preoperative Sleep Intervention on Postoperative Delirium in Infants and Toddlers Undergoing Congenital Heart Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yan Fuxia (Other)
Responsible Party: Sponsor-Investigator, Yan Fuxia, principal investigator, Chinese Academy of Medical Sciences, Fuwai Hospital
Organization: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025-2603
Record Dates: First submitted 2025-02-25; First posted 2025-03-06 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-04

CONDITIONS: Delirium - Postoperative; Sleep Problems; Congenital Heart Disease (CHD)
MeSH Terms: conditions — Emergence Delirium; Parasomnias; Heart Defects, Congenital

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Message-based bedtime routine group (Experimental): The intervention group implemented sleep hygiene education and the Message-based bedtime routine, including nutritional activities-hygiene-communication-message.
  Interventions: Behavioral: Message-based bedtime routine
- Sleep hygiene education group (Other): The control group received only sleep hygiene education.
  Interventions: Behavioral: sleep hygiene education

INTERVENTIONS:
Behavioral: Message-based bedtime routine — The intervention group implemented sleep hygiene education and the Message-based bedtime routine, including nutritional activities-hygiene-communication-message.
  Arms: Message-based bedtime routine group
Behavioral: sleep hygiene education — Sleep hygiene education includes sleep environment, sleeping location, regular sleep schedule, bedtime routines, sleeping methods, and sleeping posture.
  Arms: Sleep hygiene education group

SUMMARY:
This is a multicenter, randomized, controlled clinical trial aimed to determine whether preoperative sleep interventions could reduce the incidence of adverse outcomes, such as postoperative delirium, in sleep-disordered infants and toddlers undergoing congenital heart surgery. The study will include infants and toddlers undergoing elective cardiac surgery with sleep disorders, assessed by the Brief Infant Sleep Questionnaire (BISQ). All participants will be randomly assigned to the intervention group and Controll group in a 1:1 ratio. The intervention group received sleep hygiene education and a bedtime routine based on touch, the control group received only sleep hygiene education. The primary outcome is the incidence of postoperative delirium within 7 days after surgery or before discharge, and secondary outcomes include postoperative sleep quality, pain score, perioperative organ injury (including AKI, acute lung injury, and postoperative liver dysfunction), clinical recovery and prognosis. The results of this study will provide suggestions for the prevention of delirium after cardiac surgery.

DETAILED DESCRIPTION:
The study will be carried out in Fuwai Hospital, Chinese Academy of Medical Sciences, Anzhen Hospital Affiliated to Capital Medical University, Fuwai Central China Cardiovascular Hospital, Fuwai Cardiovascular Hospital of Yunnan Province, and Children's Hospital Affiliated to Capital Institute of Pediatrics.

The research process is as follows: Perform routine sleep disorder assessments on pediatric patients visiting the outpatient clinic. Fully inform the guardians of pediatric patients with sleep disorders of all the contents and procedures of this trial. After obtaining informed consent comprehensively and having the informed consent forms signed, conduct further assessments on the pediatric patients to determine whether they meet the inclusion and exclusion criteria. All enrolled children's guardians will receive sleep hygine education in the outpatient clinic. After stratification by research center, the random block is set to 4 - 6, the R will be used to randomly assign subjects to the experimental group and the control group at a 1:1 ratio. After randomization, the children in the experimental group receive behavioral interventions every day before surgery, specifically a bedtime routine based on massage/stroking. Guardians need to strictly implement it and cooperate with the researchers through phone calls (during the waiting period for admission) or face-to-face communication (during the preoperative hospitalization period). In the control group, parents are provided with sleep hygiene education for infants and toddlers, and no additional intervention measures are applied. To better control the quality of interventions for children aged 0 - 3 in the experimental group, the daily implementation status of parents is counted for the degree of implementation (0 - 100%) in the WeChat mini-program. Guardians record the children's daily sleep diaries (online questionnaires) before surgery. The day before surgery, they fill out the Brief Infant Sleep Questionnaire (BISQ) again and compare it with the baseline situation. After admission, children wear actigraphs until the day of surgery and until discharge after surgery to automatically record sleep-related information. After the children are enrolled in the study, relevant researchers will supervise the implementation of cognitive-behavioral interventions for the children once a day before surgery to ensure that the actigraph device functions properly during hospitalization and remind guardians to record electronic sleep diaries until the night before surgery. Follow-up will be conducted within 7 days after surgery or before discharge to evaluate outcomes such as delirium and pain. The primary outcome is the incidence of postoperative delirium, and secondary outcomes include postoperative sleep quality, pain score, perioperative organ injury (including AKI, acute lung injury, and postoperative liver dysfunction), clinical recovery and prognosis.

ELIGIBILITY:
Inclusion Criteria:

1. Age 0-3 years
2. Scheduled to undergo elective corrective surgery for congenital heart disease under cardiopulmonary bypass.
3. Children with sleep disorders who are screened by the Brief Infant Sleep Questionnaire-Revised short form (BISQ-R SF).

Exclusion Criteria:

1. Infants and toddlers who have taken any relevant preoperative treatment for sleep problems
2. The risk adjustment in congenital heart surgery-1 (RACHS-1 classification) ≥4.
3. Preoperative history of cerebral ischemia and hypoxia, developmental disorders such as autism spectrum disorders, etc.
4. Presence of any other preoperative acute or chronic medical condition (mechanical ventilation support, history of asphyxia rescue, severe hepatic or renal dysfunction, or comorbidities with other non-cardiac malformations)
5. Concurrent participation in other clinical trials
6. Refusal of the family to sign the informed consent or poor compliance of the child.

Ages: 1 Day to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 452 (Estimated)
Dates: Start 2025-04-30 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The incidence of postoperative delirium | Postoperative 7 days

SECONDARY OUTCOMES:
Mechanistic endpoint: Concentration of plasma S-100β protein | Before surgery, at the end of surgery and 24 hours after surgery
  S-100β protein was used as a surrogate biomarker for the disruption of the blood-brain barrier.
Postoperative sleep quality | Postoperative 7 days or before discharge
  Postoperative sleep quality was assessed using the Actigraph model wGT3X-BT body movement recorder. The Actigraph model wGT3X-BT was worn from the time of admission to 7 days after surgery in order to assess the sleep quality of the subjects.
Pain defined by the Face, Legs, Activity, Cry, and Consolability scale | Postoperative 7 days
  The FLACC scale is a simple and effective tool used to assess pain in infants and non-verbal patients. It stands for Face, Legs, Activity, Cry, and Consolability. Each of these five items is scored on a scale of 0 to 2, with a higher score indicating a greater degree of pain. The total FLACC score, ranging from 0 to 10, provides a quick and reliable assessment of the patient's pain level.
The incidence of postoperative Acute kidney injury | Within postoperative 7 days
The incidence of Pulmonary complication | Postoperative 7 days
The incidence of postoperative Liver dysfunction | Postoperative 7 days
Concentration of intestinal fatty acid binding protein (I-FABP) | Before surgery, at the end of surgery and 24 hours after surgery
  one of markers of intestinal injury
Concentration of zonulin | Before surgery, at the end of surgery and 24 hours after surgery
  One of markers of intestinal injury
Concentration of lipopolysaccharide (LPS) | Before surgery, at the end of surgery and 24 hours after surgery
  One of markers of intestinal injury
Concentration of lipopolysaccharide binding protein (LBP) | Before surgery, at the end of surgery and 24 hours after surgery
  One of markers of intestinal injury
Types and dosages of drugs used for postoperative sedation and analgesia | Postoperative 7 days or before discharge
Levels of inflammatory cytokines | Before surgery, at the end of surgery and 24 hours after surgery
  The inflammatory cytokines include IL-6，TNF-α，IL-1β，IFN-γ，IL-17, C-reactive protein.
Neutrophil-to-lymphocyte ratio (NLR) and Platelet-to-Lymphocyte Ratio (PLR) | Before surgery, 24 hours after surgery
  Neutrophil-to-lymphocyte ratio (NLR) and Platelet-to-Lymphocyte Ratio (PLR) are two blood biomarkers based on blood cell counts, which reflect the inflammatory and immune status of the body; they were obtained based on preoperative and postoperative blood routine tests.
The duration of postoperative mechanical ventilation | From the end of the surgery to discharge from the hospital,up to 30 days
  The total hours needing mechanical ventilation support
The length of intensive care unit stay | From the end of the surgery to discharge from the hospital,up to 30 days
  The time spent in the intensive care unit.
The length of postoperative hospital stay | From the end of the surgery to the day of discharge from the hospital,up to 30 days
Average daily cost | admission to discharge, up to 30days
  total hospitalization cost divided by total length of stay

OTHER OUTCOMES:
Long-term Sleep quality score | 30 days, 6 months, 1 year after discharge
  guardians scored sleep quality 1-5 using a sleep diary
Readmission rate | 30 days/6 months/1 year after discharge
  the rate at which a patient is readmitted to the hospital for the same or a different health problem within 30 days/six months/1 year after discharge
1-Year Mortality and Survival | 1 year after discharge
  The rate at which patients die and survive within 1 year of discharge from the hospital.

CONTACTS AND LOCATIONS:
Overall Officials: Fuxia Yan, Principal Investigator — Chinese Academy of Medical Sciences, Fuwai Hospital
Locations (1):
- Fuwai Hospital, Chinese Academy of Medical Sciences, Beijing, China

IPD SHARING:
Plan to Share IPD: No